CLINICAL TRIAL: NCT00228852
Title: Phase I/II Trial of De-Escalation of Busulfan With Fludarabine and Antithymocyte Globulin as Preparative Therapy for Hematopoietic Stem Cell Transplant for the Treatment of Severe Congenital T-Cell Immunodeficiency
Brief Title: IMM 0212: Busulfan With Fludarabine and Antithymocyte Globulin as Preparative Therapy for Hematopoietic Stem Cell Transplant for the Treatment of Severe Congenital T-Cell Immunodeficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 296-2003
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2005-09

CONDITIONS: T-Cell Immune Deficiency Diseases; Severe Combined Immunodeficiency
Keywords: Patients with severe T-cell immune deficiency diseases
MeSH Terms: conditions — Severe Combined Immunodeficiency | interventions — Busulfan; fludarabine

INTERVENTIONS:
Drug: Busulfan, Fludarabine and ATG

SUMMARY:
This is a multi-institution, single arm, non-randomized pilot study coordinated by the Pediatric Blood and Marrow Transplant Consortium. Eligible patients will have severe combined immunodeficiency syndrome (SCID) or severe T-cell immunodeficiency disorder. Patients with these disorders do not have properly functioning immune systems. Without treatment, these disorders result in early childhood death. The standard treatment used for these diseases is to give the patient a stem cell transplant from a matched donor. The donor cells can be from a family member, an unrelated marrow donor or umbilical cord blood. The donor source will impact on transplant risks and approaches to the preparative regimen.

There have been many different preparative regimens used for patients with SCIDS or severe T-cell immunodeficiency syndromes. Some patients have gotten no preparative regimen, while others have gotten only antithymocyte globulin (ATG; immune proteins made in horses that, when given, will kill lymphocytes). Still other patients have gotten conventional chemotherapy. In children treated with nothing or ATG alone, there is an increased risk of graft failure or only partial engraftment. When this happens, patients need life-long therapy with immunoglobulins to support the immune system. Children treated with chemotherapy generally have full immune recovery, but also may have major side effects from the chemotherapy. The side effects include infection, organ failure and infertility.

This protocol, in combination with a parallel study with a separate preparative regimen, will attempt to answer the question of which patients with primary immunodeficiencies need a preparative regimen and what intensity is needed. Patients will be enrolled according to disease type and donor source. The purpose of this study is to see how much chemotherapy is actually needed for the transplant to work. To be able to do this and still make the transplant work, the drugs used to temporarily weaken the immune system will be strengthened. In groups, patients will be treated with lowering doses of the busulfan to find the lowest dose of this drug that is needed to get full immune recovery. The investigators hope this regimen will result in complete immune system recovery while limiting the side effects of chemotherapy. A second purpose of this study is to track the recovery of different parts of the immune system. The investigators also want to identify whether the recovery is coming from donor stem cells or from the patient.

The patient will be admitted to the hospital to have the transplant and is expected to stay for up to 4 to 6 weeks. The preparative regimen will be made up of busulfan, fludarabine and antithymocyte globulin (ATG). After the preparative regimen, the cells from the donor will be given. To try and keep the patient's body from rejecting the donor cells and the donor cells from attacking the patient's body (graft-versus-host disease, or GVHD), cyclosporine will be given.

The investigators will draw an extra 2 - 4 teaspoons of blood at specified time points to test for immune recovery and donor cell chimerism (the portion of the blood that belongs to the donor). Standard bone marrow transplant (BMT) clinical care will be provided with respect to pretransplant evaluation, peritransplant support, and posttransplant follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following primary severe T-cell immune deficiency diseases and donor types will be eligible for this pilot trial:

  * Immunophenotype: SCIDs with decreasing T, any B, increasing natural killer (NK) with partial matched family member, unrelated donor marrow or cord blood, with or without T depletion; OR
  * Combined immunodeficiency disease (CID), including Wiskott-Aldrich and severe DiGeorge's with any donor type.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naynesh R Kamani, M.D., Study Chair — George Washington University School of Medicine
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States